CLINICAL TRIAL: NCT05466838
Title: Pancreatic Enzyme Replacement Therapy to Improve Quality of Life in Patients Undergoing Pancreaticoduodenectomy: A Pilot Randomized Controlled Trial
Brief Title: PERT to Improve Quality of Life in Patients Undergoing Pancreaticoduodenectomy: A Pilot Randomized Controlled Trial
Acronym: PERQ-UP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3962
Record Dates: First submitted 2022-06-29; First posted 2022-07-20 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Insufficiency
Keywords: Pancreaticoduodenectomy; Pancreatic enzyme replacement therapy
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PERT plus Standard of Care (Experimental): Initiation of PERT at time of discharge post pancreaticoduodenectomy with dose escalation upon symptom presentation
  Interventions: Drug: PERT at discharge; Other: Standard of Care
- Standard of Care (Other): Standard of care (no PERT) until presentation of PEI symptoms.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: PERT at discharge — Starting dose 50,000 units lipase per meal with 3 meals planned per day and 25,000 units of lipase per snack with 2 snacks planned per day. Dose escalation 100,000 units lipase with meals and 50,000 units with snacks.
  Other Names: PrCREON MINIMICROSPHERES®25 or similar (PrCotazym® ECS, PrPANCREASE® MT, PrVIOKACE™)
  Arms: PERT plus Standard of Care
Other: Standard of Care — Initiation of PERT if clinical symptoms of PEI develop or worsen. Starting dose 50,000 units lipase per meal with 3 meals planned per day and 25,000 units of lipase per snack with 2 snacks planned per day.

SUMMARY:
After pancreas surgery, patients may develop pancreatic exocrine insufficiency (PEI). PEI can be treated with oral pancreatic enzyme replacement therapy (PERT). However, the diagnosis of PEI is difficult and the guidelines about when to start PERT after pancreas surgery are conflicting. This pilot study aims to determine the feasibility of implementing a large-scale clinical trial to definitively evaluate if starting PERT immediately after surgery can improve outcomes in patients undergoing pancreas surgery.

DETAILED DESCRIPTION:
After pancreas surgery, patients may develop pancreatic exocrine insufficiency (PEI). This occurs when there are not enough exocrine cells in the pancreas to release enzymes that help with food digestion. Potential symptoms may include bloating, cramping, large and foul-smelling bowel movements (steatorrhea), and other gastrointestinal symptoms like diarrhea, weight-loss, and malnutrition. PEI can be treated with oral pancreatic enzyme replacement therapy (PERT), for example CREON. Many studies have shown that treatment of PEI with PERT is safe, effective, and may improve quality of life, reduce weight loss, improve abdominal symptoms, and may improve overall survival. However, the diagnosis of PEI is difficult and the guidelines about when to start PERT after pancreas surgery are conflicting. This pilot study aims to determine the feasibility of implementing a large-scale clinical trial to definitively evaluate if starting PERT immediately after surgery can improve outcomes in patients undergoing pancreas surgery.

Participants will be recruited from Ontario hospitals using a two-step eligibility process (pre- and post-operatively) and randomized 1:1 to receive either standard of care or PERT plus standard of care. Outcome measures will be collected 1 and 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged >18 years
2. Willing and able to provide informed consent and/or have a substitute decision maker (SDM) provide informed consent on behalf of the participant
3. Planned PD for any indication AND, at randomization
4. PD performed
5. Discharge planned within 21 days of surgery

Exclusion Criteria:

1. Contraindication to PERT including:

   1. Hypersensitivity to porcine protein, pancreatic enzymes or any excipients
   2. History of fibrosing colonopathy
   3. Unable to tolerate oral medication
2. Current use of PERT OR, at randomization
3. Use of PERT at the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients screened who consent | Baseline
  Each centre will keep a screening log of all patients who are scheduled to undergo an elective pancreaticoduodenectomy and perform pre-screening to determine eligibility. The number of eligible patients who are approached for and consent to participate, as well as the number of approached eligible patients who decline to participate (and reasons for declining) will be recorded and the proportions will be calculated
Proportion of patients screened who meet eligibility criteria | Baseline
  Each centre will keep a screening log of all patients who are scheduled to undergo an elective pancreaticoduodenectomy and perform pre-screening to determine eligibility. The eligibility criteria that are unmet will be recorded, including the additional criteria for randomization. This will be used to calculate proportions.
Adherence to PERT | 3 months
  Recorded on participant's medication tracker and calculated as a percentage of expected vs. actual doses taken.
Adherence to PERT dosing guidelines | Day 0 (Discharge)
  Review of medical record for appropriate use of PERT dosing guidelines, comparing actual prescription to dosing guideline
Adherence to PERT dosing guidelines | 1 month
  Review of medical record for appropriate use of PERT dosing guidelines, comparing actual prescription to dosing guideline
Adherence to PERT dosing guidelines | 3 months
  Review of medical record for appropriate use of PERT dosing guidelines, comparing actual prescription to dosing guideline
Completeness of dataset | 3 months
  Assessment of completeness of data, loss to follow-up and missing data and reasons for not being able to collect data
Resource requirement for definitive trial | Study completion (1.5 years)
  Each site will complete a survey at the end of the trial to report the amount of time spent on study activities

SECONDARY OUTCOMES:
Weight loss | 1 month, 3 months
  Difference in weight (kg) from baseline
Change in Digestive Symptoms Scale from Baseline | 1 month, 3 months
  Measured using PAN26 quality of life questionnaire which specific to pancreatic cancer and must be administered in conjunction with QLQ-C30. Scores range from 0 to 100 and consist of functional scales and symptoms scales. A high score on the symptoms scales indicates a high level of symptomatology. A high score on the functional scales indicates a high level of functioning.
Change in Quality of Life from Baseline | 1 month, 3 months
  Measured using the QLQ-C30 quality of life questionnaires. QLQ-C30 is a validated questionnaire that assesses health-related quality of life (QoL) in cancer patients. Scores for both questionnaires range from 0 to 100 and consist of functional scales and symptoms scales. A high score on the symptoms scales indicates a high level of symptomatology. A high score on the functional scales indicates a high level of functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Karanicolas, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (6):
- Canada (6):
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario